CLINICAL TRIAL: NCT04236128
Title: Home to Stay: an Integrated Monitoring System Using a Mobile App to Reduce Readmissions Following Colorectal Surgery
Brief Title: Home to Stay Mobile App for Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Erin Kennedy, Colorectal Surgeon (Principal Investigator), Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-0200-E
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive the same usual care as the control group plus be enrolled in the integrated discharge monitoring system.
  Interventions: Other: Mobile App
- Control Group (Active Comparator): The control group will receive usual follow up care that is currently provided at the 3 participating centres.
  Interventions: Other: Mobile App

INTERVENTIONS:
Other: Mobile App — The app will be provided to patients in hospital on post-operative day 3. On the day of discharge, the patient will be emailed a "Daily Health Check" and receive subsequent "Daily Health Check" emails on Day 1-14, 21 and 30 days following discharge. The "Daily Health Check" is a tailored questionnaire to elicit their symptoms and status of post-operative recovery. After the patient has completed the "Daily Health Check", a "Daily Health Check Summary" is emailed to the patient that summarizes their responses and provides appropriate action recommendations based on their responses ranging from: (i) suggestions for educational modules, (ii) expect a call from your health care team in the next 24 hours, (iii) call your surgeon's office today or (iv) go to the nearest emergency room. The patient's "Daily Health Check" responses are displayed in real time on a secure website that automatically "red flags" extreme responses to alert the health care team to contact the patient by telephone.

SUMMARY:
Background: Colorectal surgery includes surgery for colorectal cancer, inflammatory bowel disease and other benign diseases such as diverticulitis. In Canada, approximately 21,000 colorectal surgeries are performed each year. Patients undergoing colorectal surgery face high rates of unplanned hospital visits including readmission to hospital and Emergency Room (ER) visits. These unplanned hospital visits lead to significant distress and anxiety for patients and increased health care costs.

Research Aims: The goal is to evaluate the use of an integrated discharge monitoring system with a mobile application (app) to support colorectal surgery patients at home following discharge from hospital.

Methods: The study will include 3 hospitals across Canada. Patients will be assigned to either a control group or intervention group. Control group patients will receive standard follow up care after going home following surgery. Intervention group patients will be enrolled in an integrated discharge monitoring system using an app to monitor their progress at home following discharge after surgery. The main outcomes are to measure the number of patients with unplanned hospital visits within 30 days of discharge following surgery, the quality of patient recovery and confidence managing one's own health care. Patients are eligible if they are being discharge home after having elective colorectal surgery, are 18 years or older and speak and understand English or French. At the end of the study, the outcomes between the control group and intervention group will be compared to look for important differences.

Expected Outcomes: It is expected that the results of this study will show that the integrated discharge monitoring system will lead to a significant improvement in the quality of patient recovery and self-confidence with one's own health care, as well as significantly reduce the number of unplanned hospital visits for patients undergoing colorectal surgery in Canada.

DETAILED DESCRIPTION:
Background: Patients undergoing colorectal surgery are vulnerable during their transition from hospital to home and face high rates of unplanned hospital visits including readmission to hospital and ER visits. Not only does this lead to significant distress for patients but also translates into significant health care costs. At a patient engagement meeting with patients from across Canada led by our group, one of the main themes that emerged was the patients' sense of abandonment upon discharge from hospital following surgery. Based on this feedback, our investigative team developed and pilot tested an integrated discharge monitoring system using a mobile application (app) to support patients following discharge from hospital after colorectal surgery. The results of this pilot work provided compelling data to suggest that this integrated discharge monitoring system was feasible, highly rated by patients and may lead to a considerable decrease in 30-day unplanned hospital visits.

Research Aims: Therefore, the aim of this study is to conduct a 3 year, randomized controlled trial (RCT) to evaluate the effectiveness of an integrated discharge monitoring system to support colorectal surgery patients at home following discharge.

Methods: A RCT will be implemented at 3 high volume colorectal surgery centres across Canada. The intervention is an integrated discharge monitoring system using an app that has been developed and pilot tested in partnership with SeamlessMD. The inclusion criteria for the study are: any patient being discharged home following elective colorectal surgery, 18 years or older and able to speak and understand English or French. The primary outcome for the study is 30-day unplanned hospital visits and the secondary outcomes include patient quality of recovery and self-efficacy with one's own health care. A sample size of 670 patients is planned and will provide an 80% power to detect a 30% reduction in 30-day unplanned hospital visits, assuming a baseline 30-day unplanned hospital visit rate of 27%, 0.05 Type 1 error rate and an 80% power.

Expected Outcomes: It is expected that the results of this trial will show that the integrated discharge monitoring system leads to a significant improvement in patient satisfaction in terms of quality of recovery and self-efficacy as well as a significant reduction in 30-day unplanned hospital visits and health care costs.

ELIGIBILITY:
Inclusion Criteria:

* any patient who is being discharged to home after undergoing elective colorectal surgery
* 18 years or older
* able to speak and understand English or French
* provides informed consent

Exclusion Criteria:

* post-operative admission less than 3 days
* requiring discharge to rehabilitation centre to recover prior to being able to go home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
30-day unplanned hospital visit rate | 30 Days
  Proportion of patients who are either readmitted to any hospital or present to the ER at any hospital in the first 30 post-operative days.

SECONDARY OUTCOMES:
patient quality of recovery | 4 weeks after hospital discharge
  Quality of Recovery 15 (QoR-15) questionnaire administered to patients in both groups
patient self-efficacy to manage one's own health care | 4 weeks after hospital discharge
  Patient Activation Measure (PAM-13) administered to patients in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Erin Kennedy, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No